CLINICAL TRIAL: NCT00364273
Title: A Randomised, Double Blind, Placebo Controlled Study to Examine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetic Profile of Single Inhaled Dry Powder Doses of GSK159802 in Healthy Male Subjects
Brief Title: GSK159802 In Healthy Male Subjects And Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: B2F104300
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (14):
- Subjects receiving treatment sequence 1 : Cohort 1 (Experimental): Eligible subjects will receive placebo, GSK159802 300 micrograms, GSK159802 600 micrograms, GSK159802 900 micrograms and GSK159802 1200 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 2 : Cohort 1 (Experimental): Eligible subjects will receive GSK159802 150 micrograms, placebo, GSK159802 600 micrograms, GSK159802 900 micrograms and GSK159802 1200 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 3 : Cohort 1 (Experimental): Eligible subjects will receive GSK159802 150 micrograms, GSK159802 300 micrograms, placebo, GSK159802 900 micrograms and GSK159802 1200 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 4 : Cohort 1 (Experimental): Eligible subjects will receive GSK159802 150 micrograms, GSK159802 300 micrograms, GSK159802 600 micrograms, placebo and GSK159802 1200 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 5 : Cohort 1 (Experimental): Eligible subjects will receive GSK159802 150 micrograms, GSK159802 300 micrograms, GSK159802 600 micrograms, GSK159802 900 micrograms and placebo.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 1 : Cohort 2 (Experimental): Eligible subjects will receive placebo, salmeterol, GSK159802 low dose (LD) and GSK159802 maximum tolerated dose (MTD).
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 2 : Cohort 2 (Experimental): Eligible subjects will receive salmeterol, GSK159802 MTD, placebo and GSK159802 LD.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 3 : Cohort 2 (Experimental): Eligible subjects will receive GSK159802 LD, placebo, GSK159802 MTD and salmeterol.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 4 : Cohort 2 (Experimental): Eligible subjects will receive GSK159802 MTD, GSK159802 LD, salmeterol and placebo.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 1 : Cohort 3 (Experimental): Eligible subjects will receive placebo, salmeterol, GSK159802 300 micrograms and GSK159802 1200 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 2 : Cohort 3 (Experimental): Eligible subjects will receive salmeterol, GSK159802 1200 micrograms, placebo and GSK159802 300 micrograms.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 3 : Cohort 3 (Experimental): Eligible subjects will receive GSK159802 300 micrograms, placebo, GSK159802 1200 micrograms and salmeterol.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 4 : Cohort 3 (Experimental): Eligible subjects will receive GSK159802 1200 micrograms, GSK159802 300 micrograms, salmeterol and placebo.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol
- Subjects receiving treatment sequence 5 : Cohort 3 (Experimental): Eligible subjects will receive GSK159802 1200 micrograms, salmeterol, GSK159802 300 micrograms and placebo.
  Interventions: Drug: GSK159802; Drug: Placebo; Drug: Salmeterol

INTERVENTIONS:
Drug: GSK159802 — GSK159802 will be available with dosing strengths of 75 microgram per blister and 300 microgram per blister administered using DISKUS inhaler.
Drug: Placebo — Subjects will receive placebo administered using DISKUS inhaler.
Drug: Salmeterol — Salmeterol will be available with dosing strength of 50 micrograms per blister administered using DISKUS inhaler.

SUMMARY:
GSK159802 is a potent, inhaled, long acting selective beta-2-receptor agonist (LABA), which is being developed for once daily treatment of asthma and COPD as part of a combination product with a once daily inhaled corticosteroid and also as a standalone product for the treatment of COPD. Stimulation of the beta-2-agonist in the lung mainly relaxes bronchial smooth muscle cells which results in bronchodilation. Unwanted systemic side effects related with beta-2-agonist treatment such as tachycardia, tremor, hyperglycemia and hypokalemia are limited by local administration and also tend to show tachyphylaxis.

The LABAs that are currently available (e.g., salmeterol, formoterol) require twice-daily administration, given their duration of action. Therefore, there is significant opportunity for a once-daily inhaled medication to improve patient compliance and overall disease management by providing sustained, 24-hour bronchodilation.

ELIGIBILITY:
Inclusion criteria:

* Body mass index within the range 18.5-29.9 (kg/m2)
* Current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of < 10 pack years.

Additional criteria for Cohorts 2 and 3 only (Asthmatic Patients):

* Subjects with a documented history of mild to moderate asthma, with the exclusion of other significant pulmonary disease
* Subjects with clinically stable asthma within the 4 weeks preceding the screening visit and with a screening pre-bronchodilator FEV1 greater than 60% and less than 90% predicted.

During the screening visit, subjects must demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of > or equal to 12.0% over baseline and an absolute change of > or equal to 300 mL within 30 minutes following 400 mcg salbutamol.

Exclusion criteria:

* Any clinically relevant abnormality
* Subjects who have a screening haemoglobin values < 11 g/dL
* The subject has participated in a clinical study with a New Chemical Entity (NCE) within the past 112 days or a clinical study with any other drug during the previous 84 days
* Subjects with known hypersensitivity to salmeterol or salbutamol or any ingredients in their preparations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-08-24 (Actual); Primary Completion 2006-07-06 (Actual); Study Completion 2006-07-06 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of single inhaled doses of GSK159802. | Up to 71 days

SECONDARY OUTCOMES:
sGaw (Cohorts 1 and 2 only) and FEV1 Systemic & urine pharmacokinetics of GSK159802 and SKF-91300 Heart rate, potassium, glucose, 12-lead ECG & blood pressure | Up to 71 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study B2F104300 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/B2F104300?search=study&study_ids=B2F104300#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2F104300 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register